CLINICAL TRIAL: NCT03540459
Title: Central Apnea in Patients Receiving Ticagrelor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Les Grands Prés (Other)
Responsible Party: Principal Investigator, philippe meurin, principal investigator, Les Grands Prés
Other Study IDs: Les Grands Prés
Record Dates: First submitted 2018-05-16; First posted 2018-05-30 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: sleep polygraphy — sleep polygraphy (one night) in all included patients

SUMMARY:
all patients with a left ventricular ejection fraction superior or equal to 50% less than 2 years after an acute coronary event and receiving ticagrelor will undergo a sleep polygraphy

DETAILED DESCRIPTION:
all patients with a left ventricular ejection fraction superior or equal to 50% less than 2 years after an acute coronary event and receiving ticagrelor will undergo a sleep polygraphy the main objective of the study will be to look for central sleep apnea

ELIGIBILITY:
Inclusion Criteria:

* patient receiving ticagrelor 10 days to 2 years after an acute coronary syndrome

Exclusion Criteria:

* left ventricular ejection fraction < 50%
* patients refusal

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patient receiving ticagrelor 10 days to 2 years after an acute coronary syndrome will be included
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
central apnea index | at baseline
  mean central apnea index: apnea hypopnea index (AHI) is the scale commonly used to assess sleep disordered breathing.This scale includes central and obstructive apnea and hypopnea. The main outcome will be the central apnea index: number of central apnea per hour

SECONDARY OUTCOMES:
global apnea hypopnea index | baseline
  number of apnea and hypopnea per our

CONTACTS AND LOCATIONS:
Locations (1):
- Les Grands Prés, Villeneuve-Saint-Denis, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meurin P, Ben Driss A, Defrance C, Dumaine R, Weber H, Renaud N, Bonnevie L, Mouram S, Tabet JY. Central sleep apnea after acute coronary syndrome and association with ticagrelor use. Sleep Med. 2021 Apr;80:39-45. doi: 10.1016/j.sleep.2021.01.026. Epub 2021 Jan 20. PMID 33550173